CLINICAL TRIAL: NCT05182424
Title: Randomized Controlled Trial of the Myndlift BPT App
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: New York University (Other)
Collaborators: Myndlift Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2022-5839
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-11

CONDITIONS: ADHD; Behavioral Disorder
Keywords: ADHD; Behavioral Disorder; Telehealth; Behavioral Parent Training (BPT); Parents; Parent; Parent Training; Children; Disruptive Behaviors
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Mental Disorders; Problem Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myndlift BPT Immediate Treatment (Experimental): After the completion of consent, a battery of baseline assessments will be completed by the parent. Children will not be involved in the study assessment or interventions-only parents/caregivers. Parent(s) will be emailed baseline and post-treatment assessment surveys through Qualtrics to complete. Following completion of baseline assessment, study staff will meet with the parent via Zoom to review any questions with the consent and review and discuss questions/issues with the baseline assessment. Following completion of the post-treatment assessment, study staff will meet with the parent via Zoom to review and discuss questions/issues with the post-treatment assessment. Following this review, the post-treatment interview will be completed. Having study staff present has been found useful by parents should they have any questions or concerns about items on surveys.
  Interventions: Behavioral: Myndlift BPT App & As-Needed Therapist Support
- Waitlist Control Group (Other): Following completion of consent and baseline assessment, parent participants randomly assigned to the waitlist condition will be requested to wait for a period of 12 weeks before accessing the program, modules, and receiving therapist support. They will be required to answer the time 2 (at 12 weeks following completion of the baseline assessment) assessment prior to starting the process. The time 2 assessment for the waitlist condition is identical to the post-treatment assessment for participants in the Myndlift BPT group except that questions related to experience with Myndlift BPT will not be included.
  Interventions: Behavioral: Myndlift BPT App & As-Needed Therapist Support

INTERVENTIONS:
Behavioral: Myndlift BPT App & As-Needed Therapist Support — BPT is based on social learning and operant conditioning principles in which parents are instructed to utilize methods to facilitate positive behaviors in their child and reduce challenging behaviors. Myndlift BPT translates established content and processes into a digital format to be delivered through a mobile app. Myndlift content consists of 10 components, designed to be completed in a self-directed manner by parents, over the course of approximately 10 weeks (total weeks depends upon parent's pace through the program).
  In this project, trained and supervised doctoral- and masters-level students will serve as study therapists and meet with parents via a secured, password-protected Zoom platform to introduce parents to the Myndlift BPT (first session before start of the BPT), to support and problem solve BPT skills acquisition (during the Myndlift BPT), and at the end of the Myndlift BPT (to review the intervention content and consider the maintenance of skills).

SUMMARY:
We propose addressing these aims by conducting a randomized controlled trial (RCT) that will evaluate the hybrid BPT (Myndlift BPT) compared to a wait-list control group. All participants will receive the Myndlift BPT at either the initial point of randomization or following the wait-list time period.

The Myndlift BPT consists of 10, self-directed app-based BPT modules accessible through an online mobile application with each module requiring up to 30 minutes of parent's time. Therapist contact ("parent-therapist consults") will be based on parent need. We anticipate approximately six standard 20-minute therapist contacts during the Myndlift BPT (one prior to the start of the app-based BPT modules, four parent-therapist consults during the app-based BPT modules, and one final parent-therapist consult at the end of app-based BPT modules). Additional parent-therapist consults will be based on parents' needs. In addition, therapists will monitor parent progress and challenges with the app-based BPT modules using a web-based therapist portal. The therapist may initiate additional parent-therapist consults if s/he deems it necessary based on client progress, and contacts can be longer than 20 minutes if needed. All consults are completed through Zoom telehealth platform.

Given the self-directed nature of the Myndlift BPT (parents decide how frequently they access the app-based modules of BPT and practice the skills), parent involvement in the intervention will vary slightly in duration. However, based on the literature and routine practice, we anticipate parents completing one module/week in the app-based parent feature for a total of 10 weeks with an additional therapist supported session at the start of the intervention and one at the end of the intervention for a total of 12 weeks of involvement in the Myndlift BPT. The research assessment (see details below) will occur at baseline and at the end of Myndlift BPT. Given that the assessments are linked to participant progress in the Myndlift BPT, participant involvement in the study will also slightly vary, but we anticipate that most parents will complete the assessment during a standard 12-week Myndlift BPT schedule.

DETAILED DESCRIPTION:
Over the past several decades, much of the literature on attention-deficit/hyperactivity disorder (ADHD) and other disruptive behavior disorders (DBDs; i.e., conduct disorder/CD and oppositional defiant disorder/ODD) in children has focused on evaluating the effectiveness of different treatment approaches. While research has determined that pharmacological treatments can be considered well-established and evidence-based, they are not always sufficient - in that, a variety of individual differences may limit the effectiveness of drug treatment for any given individual - and can lead to a host of undesired side effects (Chacko et al., 2015). Additionally, parents are often resistant to medicating their children, particularly at younger ages, and prefer to engage in other treatment options, when possible (Charach et al., 2006). Research on psychosocial approaches has likewise determined that behavioral parent training (BPT) interventions are well-established and evidence-based, and over time, BPT has become one of the most well-studied and efficacious psychosocial interventions for families with children with ADHD (Chacko et al., 2015).

In light of the growing importance of readily available and accessible hybrid (online, self-directed with therapist support) BPT, our research team, in collaboration with Myndlift (a leading technology-based company that translates evidence-based non-pharmacological interventions into online delivery formats), proposes a study of hybrid BPT for parents of children with or at risk for ADHD. The specific aims of the study are: 1) to determine the feasibility and acceptability/satisfaction with the hybrid BPT and, 2) relative to a wait-list control condition, to determine the impact of the hybrid BPT on child (ADHD and related behavioral problems; impairment) and parent (parenting behavior, parental stress, parenting competence) outcomes.

We propose addressing these aims by conducting a randomized controlled trial (RCT) that will evaluate the hybrid BPT (Myndlift BPT) compared to a wait-list control group. All participants will receive the Myndlift BPT at either the initial point of randomization or following the wait-list time period.

The Myndlift BPT consists of 10, self-directed app-based BPT modules accessible through an online mobile application with each module requiring up to 30 minutes of parent's time. Therapist contact ("parent-therapist consults") will be based on parent need. We anticipate approximately six standard 20-minute therapist contacts during the Myndlift BPT (one prior to the start of the app-based BPT modules, four parent-therapist consults during the app-based BPT modules, and one final parent-therapist consult at the end of app-based BPT modules). Additional parent-therapist consults will be based on parents' needs. In addition, therapists will monitor parent progress and challenges with the app-based BPT modules using a web-based therapist portal. The therapist may initiate additional parent-therapist consults if s/he deems it necessary based on client progress, and contacts can be longer than 20 minutes if needed. All consults are completed through Zoom telehealth platform.

Given the self-directed nature of the Myndlift BPT (parents decide how frequently they access the app-based modules of BPT and practice the skills), parent involvement in the intervention will vary slightly in duration. However, based on the literature and routine practice, we anticipate parents completing one module/week in the app-based parent feature for a total of 10 weeks with an additional therapist supported session at the start of the intervention and one at the end of the intervention for a total of 12 weeks of involvement in the Myndlift BPT. The research assessment (see details below) will occur at baseline and at the end of Myndlift BPT. Given that the assessments are linked to participant progress in the Myndlift BPT, participant involvement in the study will also slightly vary, but we anticipate that most parents will complete the assessment during a standard 12-week Myndlift BPT schedule.

ELIGIBILITY:
Inclusion Criteria:

* the child must be between the ages of 3-11 at the time of baseline/pretreatment data collection;
* the child must have an elevated score based on parent-report on the Inattention and/or Hyperactivity/Impulsivity Symptom Index of the ADHD Rating Scale- 5 (Dupual et al., 2016)
* the parent/caregiver must be a fluent English speaker;
* the parent/caregiver must be the legal guardians of and have full-time child care responsibilities for their child (parents/caregiver with limited contact with their child will not have the opportunity to sufficiently practice the BPT skills),
* the parent/caregiver must have reliable and stable mobile internet access,
* the parent/caregiver must use an Apple iOS operating system (Myndlift BPT is only available in iOS 9 or above) the parent/caregiver and their child must reside in the United States.

Exclusion Criteria:

* the child or parent/caregiver presents with emergency psychiatric needs that require services beyond those that can be managed within this intervention format (e.g., hospitalization, specialized placement outside the home); In this case, an active intervention by research staff to secure what is needed will be made;
* if the child has an elevated score for Autism Spectrum Disorder on the Developmental Behavior Checklist-Autism Screening Algorithm (youth with ASD often require considerably more intervention; and,
* if the parent/caregiver is currently enrolled or has recently enrolled in any type of BPT program (i.e., past two years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in ADHD Rating Scale-5: Home Version (ADHD-RS5) from Baseline to 12-week Follow up | Baseline, 12 Week Follow Up
  The ADHD-RS5 Home Version is a rating scale based on the diagnostic criteria for ADHD as described in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). The ADHD-RS5 consists of two symptom subscales: Inattention (9 items) and Hyperactivity-Impulsivity (9 items), as well as a Total Scale (18 items). In addition, the ADHD Rating Scale-5 assesses six domains of impairment that are common among children with ADHD: relationships with significant others (family members for the home version and teachers for the school version), peer relationships, academic functioning, behavioral functioning, homework performance, and self-esteem. When using the ADHD Rating Scale-5, respondents complete each set of impairment items twice, first after rating the inattention symptom items and again after rating the hyperactivity-impulsivity items.
Change in Disruptive Behavior Disorders (DBD) Rating Scale from Baseline to 12-week Follow up | Baseline, 12 Week Follow Up
  The DBD scale is a 45-item measure that asks parents to rate symptoms of ADHD, ODD, and CD on a 4-point Likert scale (i.e., "not at all", "just a little", "pretty much", or "very much"), with higher scores indicating more problems. For this study, the average scores for the DSM ODD and CD will be used.
  Support for the scale's reliability and validity have been reported in past samples, with acceptable levels of internal consistency (.82) and concurrent correlations with other measures used for diagnosis of ADHD and ODD being reported (Pelham et al., 2005).
Change in Impairment Rating Scale - Parent/Teacher Version (IRS) from Baseline to 12-week Follow up | Baseline, 12 Week Follow Up
  The IRS is a multidimensional measure that assesses functioning across domains. Specifically, the IRS qualifies and quantifies impairment present in a child's life, both in school and non-school settings. The scale has parent and teacher versions that ask about the degree to which the child has problems that warrant treatment, intervention, or special services in specific areas of functioning. For children ages 4 through 12, the IRS has shown good psychometric properties and has empirically derived cutoff points.
  The IRS asks the informant to respond using a 7-point scale that ranges from "No problem; definitely does not need treatment or special services" to "Extreme problem; definitely needs treatment or special services." The IRS exhibits concurrent, discriminant, and convergent validity, and acceptable levels of temporal stability.
Change in Parenting Stress Index - Short Form (PSI-SF) from Baseline to 12-week Follow up | Baseline, 12 Week Follow Up
  The PSI-SF measures the level of stress in the parent-child relationship and is appropriate for use with children aged 1 month to 12 years. It was derived from the longer Parenting Stress Index and consists of 36 statements, each rated on a 1 to 5 scale (1=strongly disagree, 5=strongly agree), which produces a Total Stress score. The items also cluster to produce three subscale scores (Parental Distress, Difficult Child, and Parent-child Dysfunctional Interaction) each derived from ratings of 12 items.
Change in The Parenting Scale (PS) from Baseline to 12-week Follow up | Baseline, 12 Week Follow Up
  The PS is a 30-item parent self-report measure of dysfunctional parenting in discipline situations. For each item, parents are asked to rate on a seven-point Likert scale about their likelihood of using a specific discipline strategy. It yields a total score based on three factors: Laxness (permissive discipline), Overreactivity (authoritarian discipline, displays of anger, meanness, and irritability), and Verbosity
  MYNDLIFT BPT SURVEY PACKET 8
  (overly long reprimands or reliance on talking). The total score has demonstrated adequate internal consistency (α = .84) and good test-retest reliability (r = .84).
Change in Parenting Sense of Competence (PSOC) from Baseline to 12-week Follow up | Baseline, 12 Week Follow Up
  The Parenting Sense of Competence (PSOC) scale is a commonly used measure of parental self-efficacy. The PSOC is a 17-item questionnaire that measures overall parenting sense of competence and includes two sub-scales measuring parental satisfaction and parental self-efficacy. The Efficacy factor examines the parents' competence, capability levels, and problem-solving abilities in their parental role; the Satisfaction factor examines the parents' anxiety, motivation, and frustration.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Chacko, PhD, Principal Investigator — New York University
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No